CLINICAL TRIAL: NCT03701711
Title: A Phase I Study of Lenalidomide in Combination with Dexamethasone in Anti-MAG Demyelinating Sensorimotor Neuropathy
Brief Title: Lenalidomide in Anti-MAG Neuropathy: Phase 1b Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Higher than expected occurrence of VTE (venous thromboembolic event)
Sponsor: Ohio State University (Other)
Collaborators: Celgene Corporation (Industry); University of Michigan (Other)
Responsible Party: Principal Investigator, Bakri Elsheikh, Professor of Neurology, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018H0150
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-03

CONDITIONS: Demyelinating Sensorimotor Neuropathy
Keywords: Lenalidomide
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Intervention Model Description: Single arm dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenalidomide escalation and expansion (Experimental): Among the participants who will be receiving lenalidomide, the first 12 participants will be in the dose escalation phase; with the subsequent 8 participants anticipated to receive dose expansion.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Dose Escalation
  Patients in the dose escalation phase will receive oral treatment with:
  Lenalidomide: 10, 15, or 25 mg on Days 1-21 of every 28-day cycle Dexamethasone: 20mg on Days 1,8,15 and 22
  Starting doses of Lenalidomide will be assigned at the time of registration.
  Dose Expansion
  Once the MTD has been established or determined, 8 additional patients will be treated at the MTD of lenalidomide at the same schedule as above. Dexamethasone will be given at the same dose as in the dose escalation portion of the study.
  Other Names: Revlimid

SUMMARY:
Anti-myelin-associated glycoprotein (MAG) is a rare autoimmune disorder of the peripheral nerves that presents with weakness, gait imbalance, and loss of sensation. It almost always occurs in the setting of excess protein buildup in the body in the form of immunoglobulin monoclonal (IgM) gammopathy. Anti-MAG neuropathy currently has no established therapies. It is diagnosed through blood tests (anti-MAG and IgM), nerve conduction studies (which showed marked velocity slowing), and clinical exam findings.The efficacy of lenalidomide has been demonstrated in anti-MAG peripheral neuropathy with two separate dosing regimens: 25mg on days 1-21 of each 28 day cycle in conjunction with oral dexamethasone 20mg/day on days 1-4 of each cycle as well as at 5mg on days 1-21 of each cycle without oral dexamethasone. This phase 1 study aims to determine the maximum tolerated dose (MTD) of Lenalidomide in patients with anti-MAG neuropathy. We will explore preliminary efficacy and postulate that this drug is effective in this subset of patients, using preselected, specifically tailored outcome measures that encompass quality of life, neurologic function, serum protein levels, and focused measures of proprioception.

DETAILED DESCRIPTION:
Primary Objective

1. To determine the maximum tolerated dose (MTD) in phase I of lenalidomide and recommended dose in an extension cohort of lenalidomide of anti-MAG patients
2. To examine the safety profile of lenalidomide in anti-MAG patients Secondary Objective To explore preliminary efficacy by using preselected, specifically tailored outcome measures that encompass quality of life, neurologic function, serum protein levels, and focused measures of proprioception

Study Design Part 1: Dose Escalation

Patients in the dose escalation phase will receive oral treatment with:

Lenalidomide: 10, 15, or 25 mg on Days 1-21 of every 28-day cycle Dexamethasone: 20mg on Days 1,8,15 and 22

Starting doses of Lenalidomide will be assigned at the time of registration.

To find the MTD and select the dose level for each cohort enrolled, we will use the Bayesian optimal interval design (BOIN).3-4 BOIN is implemented in a way that is similar to the traditional 3+3 design but has superior operating characteristics that are comparable to much more complex model-based designs, like the continual reassessment method (CRM).

The target toxicity rate will be 0.3 and the maximum sample size will be 12 patients. The BOIN design does not require a fixed cohort size throughout the trial. Thus, we will initially enroll in cohorts of size 1 but can modify subsequent cohort sizes as desired.

After the enrollment of the maximum sample size, the MTD will be selected using isotonic regression. The MTD will be the dose with the estimated toxicity rate closest to the target rate of 0.3.

Part 2: Dose Expansion

Once the MTD has been established or determined, 8 additional patients will be treated at the MTD of lenalidomide at the same schedule as above. Dexamethasone will be given at the same dose as in the dose escalation portion of the study.

Patients who have not had disease progression, have experienced acceptable toxicity or have not withdrawn for any other reason after 24 months will be eligible to continue protocol treatment at their current dose level until disease progression, unacceptable toxicity, or refusal. Those patients who have not progressed and who have experienced unacceptable toxicity may be eligible for re-treatment at a lower dose. A maximum of 2 reductions are allowed.

Criteria for discontinuation of protocol therapy include:

* Request by the patient to withdraw
* Unacceptable adverse events
* Treatment delay of >4weeks
* Intercurrent illness which would, in the judgment of the investigator, affect assessments of clinical status to a significant degree that require discontinuation of drug
* Non-protocol chemotherapy, or an experimental drug during the trial

Patients who discontinue treatment for any of the above reasons will go to event monitoring. Once a patient has entered the event monitoring phase of the trial, his/her therapy is at the discretion of the treating physician. Patients' charts will be reviewed for progression and survival endpoints during visits with treating physicians.

Peripheral blood (10ml purple top EDTA for immediate analysis and 6ml red top for possible later cytokine evaluation) will be collected at pre-treatment and after cycles 1,2,3,6,9,12, as well as 18 and 24 (for extension phase) for immunome correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have an Anti-Myelin Associated Glycoprotein titer

  * Patients must have Distal acquired demyelinating sensorimotor (DADS) peripheral neuropathy phenotype as defined per European Federation of Neurological Societies (EFNS) demyelinating criteria with preferential distal nerve involvement, as captured per terminal latency index [terminal distance/(conduction velocity x terminal latency)], in the setting of a monoclonal gammopathy
  * Patients must be at least 18 years of age with no evidence of multiple myeloma, light chain amyloidosis or other hematologic disorder requiring treatment.
  * Patient may be enrolled at any time from last line of therapy.
  * Patients must have ANC > 1000/µL and Platelets ≥75,000/µL
  * Patients must have adequate hepatic function as evidenced by: total bilirubin < 1.5 mg/dL, alkaline phosphatase < 3X the ULN, and AST/ALT < 2X the ULN.
  * Patients must be able to take any of the following once lenalidomide starts and for at least 5 days after last dose lenalidomide: 1) 81-325 mg of coated aspirin daily; 2) full dose warfarin (target INR 2-3); 3) 2.5 mg or above of apixaban twice daily; 4) low molecular weight heparin; 5) 20 mg or above of rivaroxaban daily.
  * Patients must have adequate renal function as evidenced by serum creatinine < 2mg/dL or calculated creatinine clearance of ≥ 40ml/min within 14 days of registration using MDRD formula.
  * Patient must be able to swallow capsule or tablet.
  * Patients must provide informed consent.
  * All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
  * Two negative pregnancy tests will be required for all women of child bearing potential, with the second negative test having been at least 7 days prior to starting the study drug. Breast feeding is not permitted.
  * Fertility requirements

    * Female patients with child bearing potential must have two negative pregnancy tests, with the second negative test having been at least 7 days prior to starting the study drug.
    * Male patients must agree to use an adequate method of contraception starting from screening to 90 days after stopping the drug.
    * Female patients must be either posy-menopausal, free from menses ≥2 yrs., surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from sexual activity starting from screening to 90 days after stopping the drug.
    * Female patients of child bearing potential must agree to comply with the fertility and pregnancy test requirements dictated by the Rev-Assist program.

Exclusion Criteria:

* • Patient with concurrent hematologic or oncologic malignancy requiring systemic treatment

  * History of allergic reaction (including erythema nodosum) to lenalidomide
  * Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from the side-effects of surgery
  * Patients with a history of gastrointestinal surgery or other procedure that might, in the opinion of the investigator(s), interfere with the absorption or swallowing of the study drugs.
  * Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to them by the study staff.
  * Any other medical condition, including mental illness or substance abuse deemed by the investigator(s) to likely interfere with the patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
MTD | Treatment duration up to 24 months
  the maximum tolerated dose (MTD) of lenalidomide

SECONDARY OUTCOMES:
Dose Extension | Treatment duration up to 24 months
  the recommended dose extension; subsequent to the maximum tolerated dose (MTD) of lenalidomide

OTHER OUTCOMES:
EQ-5D-5L | Treatment duration up to 24 months
  A self-reported descriptive system that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems(2), moderate problems(3), severe problems(4) and extreme problems(5). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The new version can define 3,125 (=55) different health states. The five figure score represents a 1-5 score in each of 5 domains; the lower the score in each domain the less severe the problems in that domain.
Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | Treatment duration up to 24 months
  The INCAT (Inflammatory Neuropathy Cause and Treatment) disability score is a measure of activity limitation. It is used frequently as a primary endpoint in inflammatory polyneuropathy clinical trials. The INCAT disability score combines arm and leg disability in a total score ranging from 0 (no signs of disability) to 12 (most severe disability score). It provides a good functional description of the arms and legs in a checklist form suitable for interviewing patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bakri Elsheikh, MBBS, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Stino AM, Bumma N, Smith R, Davalos L, Allen J, Ye JC, Pianko M, Campagnaro E, Fierro C, Awad A, Murdock B, Pietrzak M, Loszanski G, Kline DM, Efebera Y, Elsheikh B. Lenalidomide in the treatment of anti-myelin-associated glycoprotein neuropathy: A phase 1 study to identify the maximum tolerated dose. Eur J Neurol. 2024 Mar;31(3):e16164. doi: 10.1111/ene.16164. Epub 2023 Nov 28. PMID 38015467